CLINICAL TRIAL: NCT00479063
Title: Modic Changes Are Not Associated With a Higher Risk of Chronic Low Back Pain Among Southern European Subjects. A Case Control Study
Brief Title: Association of Lumbar MODIC Changes With Chronic Low Back Pain in Southern European Subjects
Acronym: MODIC 2
Status: Completed | Type: Observational
Sponsor: Kovacs Foundation (Other)
Responsible Party: Francisco M. Kovacs, Director of Scientific Department, Kovacs Foundation
Other Study IDs: FK-R-16
Record Dates: First submitted 2007-05-24; First posted 2007-05-25 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Low Back Pain
Keywords: MODIC changes; chronic low back pain; magnetic resonance imaging (MRI); vertebrae; intervertebral disc
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cases: All subjects screened for this study were aged 30 to 50 years, had been referred to participating Radiology services, and underwent a lumbar MRI. Cases had been referred for a lumbar MRI for LBP lasting > 90 days.
- Controls: All subjects screened for this study were aged 30 to 50 years, had been referred to participating Radiology services, and underwent a lumbar MRI. Controls were headache patients who had been referred for a cranial MRI, which turned out to be normal, and who either had no history of LBP or had only experienced one episode in their life, which had lasted for less than 7 days.

SUMMARY:
In this case-control study, cases were chronic LBP patients aged 30-50 in whom a lumbar MRI had been prescribed. Controls were subjects aged 30-50 in whom a cranial MRI had been prescribed for headache, who did not suffer from LBP and had no history of clinically relevant LBP. Two hundred and forty cases and 64 controls were recruited consecutively in Radiology services across six cities in Spain. Imaging findings and subjects' characteristics were gathered through previously validated instruments. Radiologists who interpreted MRIs were blinded to subjects' characteristics. A multivariate logistic regression model was developed to assess the association of Modic changes with LBP, adjusting for sex, age, body-mass index, lifetime exposure to smoking, physical activity, and disk degeneration.

ELIGIBILITY:
Inclusion Criteria:

* For all subjects: age between 35 and 50 years.
* For subjects with LBP: having a diagnosis of chronic low back pain (of 3 or more months' duration) as the reason for an MRI.
* For subjects without LBP: subjects with a cranial MRI (described as normal) for cephalalgia, and who had neither current LBP nor history of LBP.

Exclusion criteria were: history of spine surgery, current pregnancy, scoliosis with >15º curvature, vertebral fractures, "red flags" for potential underlying systemic diseases (oncologic disease during the previous 5 years, constitutional symptoms -unexplained weight loss, fever, chills-, history of intravenous drug use, or immunocompromised host), or signs suggesting cauda equine syndrome (relevant or progressive paresia, loss of sphincter control or saddle anesthesia).

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Cases: chronic LBP patients aged 30-50 in whom a lumbar MRI had been prescribed. Controls: subjects aged 30-50 in whom a cranial MRI had been prescribed for headache, who did not suffer from LBP and had no history of clinically relevant LBP.
Sampling Method: Non-Probability Sample
Enrollment: 304 (Actual)
Dates: Start 2010-02; Primary Completion 2010-12 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco M Kovacs, MD, PhD, Study Director — Kovacs Foundation, Palma de Mallorca, Spain; Carlos Campillo, MD, Principal Investigator — IbSalut, Palma de Mallorca, Spain
Locations (1):
- Kovacs Foundation, Palma de Mallorca, Balearic Islands, Spain

REFERENCES:
- [Background] Modic MT, Steinberg PM, Ross JS, Masaryk TJ, Carter JR. Degenerative disk disease: assessment of changes in vertebral body marrow with MR imaging. Radiology. 1988 Jan;166(1 Pt 1):193-9. doi: 10.1148/radiology.166.1.3336678.
- [Background] Toyone T, Takahashi K, Kitahara H, Yamagata M, Murakami M, Moriya H. Vertebral bone-marrow changes in degenerative lumbar disc disease. An MRI study of 74 patients with low back pain. J Bone Joint Surg Br. 1994 Sep;76(5):757-64. PMID 8083266
- [Background] Stirling A, Worthington T, Rafiq M, Lambert PA, Elliott TS. Association between sciatica and Propionibacterium acnes. Lancet. 2001 Jun 23;357(9273):2024-5. doi: 10.1016/S0140-6736(00)05109-6. No abstract available. PMID 11438138